CLINICAL TRIAL: NCT06194812
Title: Evaluation of the Responsibility and Minimal Clinical Important Change of the Turkish Versions of the Fear-Avoidance Beliefs Questionnaire, Tampa Kinesiophobia Scale,and Pain Catastrophizing Scale in Patients With Chronic Neck Pain.
Brief Title: Minimal Clinical Important Change of the Turkish Versions of the FABQ TKS, and PCS in Patients With Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Irmak ÇAVUŞOĞLU, Assistant professor, Acibadem University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-19/651
Record Dates: First submitted 2023-12-13; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Neck Pain; Kinesiophobia; Fear of Movement
MeSH Terms: conditions — Neck Pain; Kinesiophobia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- İNTERVENTİON (Other): The surveys in the study will be applied to the patients in this group and initial and final measurements will be taken.
  Interventions: Other: Pain Catastrophizing scale

INTERVENTIONS:
Other: Pain Catastrophizing scale — Participants' fear and avoidance behaviors will be evaluated with the Fear Avoidance Beliefs Questionnaire (KKBS) (Appendix 2).
  Participants' fear of movement will be evaluated with the Tampa Kinesiophobia Scale (TKS) (Appendix 3).
  Pain Catastrophizing Scale (PAS) (Appendix 4) will be used to evaluate the participants' pain-related thoughts and feelings.
  The amount of improvement in symptoms perceived by the participants will be evaluated at the end of the treatment with the Global Perceived Impact Scale (GAES) (Appendix 5). Participants were asked "How would you describe your current situation compared to the beginning of treatment?" question will be asked.
  Other Names: Fear-Avoidance Beliefs Questionnaire, and Pain Catastrophizing scale; Tampa Kinesiophobia scale

SUMMARY:
To investigate the reliability and sensitivity of the Fear-Avoidance Beliefs Questionnaire, Tampa Kinesiophobia Scale, and Pain Catastrophizing Scale in patients with chronic nonspecific neck pain undergoing multidisciplinary rehabilitation and to determine the most appropriate minimally clinically significant difference values in order to increase confidence in their use in clinical practice and research for this patient population. Therefore, the current study aims to evaluate the answerability and minimal clinical significance of the Turkish versions of the Fear-Avoidance Beliefs Questionnaire, Tampa Kinesiophobia scale, and Pain Catastrophizing scales in patients with non-specific chronic neck pain.

DETAILED DESCRIPTION:
To investigate the reliability and sensitivity of the Fear-Avoidance Beliefs Questionnaire, Tampa Kinesiophobia Scale, and Pain Catastrophizing Scale in patients with chronic nonspecific neck pain undergoing multidisciplinary rehabilitation and to determine the most appropriate minimally clinically significant difference values in order to increase confidence in their use in clinical practice and research for this patient population. Therefore, the current study aims to evaluate the answerability and minimal clinical significance of the Turkish versions of the Fear-Avoidance Beliefs Questionnaire, Tampa Kinesiophobia scale, and Pain Catastrophizing scales in patients with non-specific chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:A definitive diagnosis of chronic nonspecific neck pain (documented history of neck pain lasting more than twelve weeks without a recognizable, specific pathoanatomical cause of the pain)

* Good Turkish communication skills
* Both genders must be between the ages of 18 and 65,
* Agreeing to participate in the research and signing the voluntary consent form

Exclusion Criteria:

* Systemic disease, cognitive impairment (Mini Mental State Examination <24),

  * Recent (<12 weeks) myocardial infarction, cerebrovascular accident
  * Rheumatoid arthritis, neurological disorders, radiculopathy, infection, tumor, osteoporosis, vertebral fracture, trauma and surgery in the cervical region.
  * Having previously received any exercise therapy and/or pain neuroscience training.
  * Refusal of treatment or failure to comply with treatment (

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Fear-Avoidance | baseline and after 8 weeks
  It is aimed to evaluate the responsibility and minimal clinical significance of the Fear-Avoidance Beliefs Questionnaire in patients with non-specific chronic neck pain.

SECONDARY OUTCOMES:
Kinesiophobia | baseline and after 8 weeks
  It is aimed to evaluate the responsibility and minimal clinical significance of the Turkish versions of the Tampa Kinesiophobia scale in patients with non-specific chronic neck pain.
Pain Catastrophizing | baseline and after 8 weeks
  It is aimed to evaluate the responsibility and minimal clinical significance of the Turkish versions of the Pain Catastrophizing scale in patients with non-specific chronic neck pain.

CONTACTS AND LOCATIONS:
Overall Officials: Nuray Alaca, assoc.prof., Study Chair — Acibadem University; Elif Esma Safran, PhD, Study Chair — Acibadem University
Locations (1):
- Avicenna Hospital, Istanbul, Turkey (Türkiye)